CLINICAL TRIAL: NCT02222233
Title: Relative Bioavailability of Single Doses of 200 mg BI 671800 HEA Administered Orally as a Delayed Release (Enteric Coated) Tablet; or Via the EnterionTM Capsule as Solution to the Jejunum, Ascending Colon or Descending Colon; or Via the EnterionTM Capsule as Particulate to the Ascending Colon. An Open-label, Five Periods, Fixed Sequence Phase I Study in Healthy Male Volunteers
Brief Title: Relative Bioavailability of BI 671800 HEA in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1268.60
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets

ARMS (5):
- BI 671800 HEA delayed release (enteric coated) tablet (Experimental)
  Interventions: Drug: BI 671800 HEA delayed release (enteric coated) tablet
- BI 671800 HEA solution released in jejunum (Experimental): BI 671800 HEA solution in the Enterion® capsule released in the jejunum
  Interventions: Drug: BI 671800 HEA solution
- BI 671800 HEA solution released in ascending colon (Experimental): BI 671800 HEA solution in the Enterion® capsule released in the ascending colon
  Interventions: Drug: BI 671800 HEA solution
- BI 671800 HEA solution released in descending colon (Experimental): BI 671800 HEA solution in the Enterion® capsule released in the descending colon
  Interventions: Drug: BI 671800 HEA solution
- BI 671800 HEA particulate released in ascending colon (Experimental): BI 671800 HEA as particulate in the Enterion® capsule released in the ascending colon
  Interventions: Drug: BI 671800 HEA particulate

INTERVENTIONS:
Drug: BI 671800 HEA delayed release (enteric coated) tablet
  Arms: BI 671800 HEA delayed release (enteric coated) tablet
Drug: BI 671800 HEA solution
  Arms: BI 671800 HEA solution released in ascending colon; BI 671800 HEA solution released in descending colon; BI 671800 HEA solution released in jejunum
Drug: BI 671800 HEA particulate
  Arms: BI 671800 HEA particulate released in ascending colon

SUMMARY:
To determine the relative bioavailability of single doses of 200 mg BI 671800 HEA (choline) administered as a delayed release (enteric coated) tablet; or via the EnterionTM capsule as solution to the jejunum, ascending or descending colon, or as particulate to the ascending colon

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males subjects
2. Aged 21-65 years
3. Body Mass Index (BMI) of 18.5-29.9 kg/m2 inclusive
4. Subjects must demonstrate their ability to swallow an empty size 000 capsule
5. Must be willing and able to participate in the whole study and must provide written informed consent

Exclusion Criteria:

1. Participation in a clinical research study involving investigational drugs or dosage forms within the previous 3 months
2. Subjects who have previously been enrolled in this study
3. Subjects who have ever sought advice from or been referred to a general practitioner or counsellor for abuse or misuse of alcohol, non medical drugs, medicinal drugs or other substance abuse e.g. solvents
4. Subjects who admit to any current or previous use of Class A drugs such as opiates, cocaine, ecstasy, lysergic acid diethylamide (LSD) and intravenous amphetamines (Subjects who admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs of abuse test and have been abstinent for at least 12 months)
5. Positive drugs of abuse test result
6. Regular alcohol consumption >21 units per week (1 Unit = ½ pint beer, a 25 mL shot of 40% spirit or a 125 mL glass of wine)
7. Current smokers and those who have smoked within the last 6 months. A breath carbon monoxide reading of greater than 10 ppm at screening
8. Radiation exposure from clinical trials, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 millisievert (mSv) in the last twelve months or 10 mSv in the last five years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.
9. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the Investigator, repeated alanine aminotransferase (ALT), aspartame aminotransferase (AST), gamma-glutamyltransferase (GGT), alkaline phosphatase (ALP) or Total bilirubin above upper limit normal (ULN)
10. History of gastrointestinal surgery (with the exception of appendectomy unless it was performed within the previous 12 months)
11. History of clinically significant disease such as cardiovascular, renal, hepatic, respiratory, central nervous system (CNS), metabolic and particularly gastrointestinal disease, especially peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's Disease or Irritable Bowel Syndrome
12. History of adverse reaction or allergy to study drug or its excipients, e.g. lactose or rescue medication (if specified by the Sponsor). If subject suffers from hayfever they must not have or be expecting to have symptoms during the study period
13. Acute diarrhoea or constipation in the 7 days before the predicted first study day. If screening occurs >7 days before the first study day, this criterion will be determined on first study day. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than three times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day
14. Donation of blood or significant blood loss within the previous three months
15. Presence of non-removable metal objects such as metal plates, screws, etc, in the abdominal region of the body (with the exception of sterilisation clips)
16. Subjects will be excluded from the study if they are considered by the Investigator to be at risk of transmitting, through blood or other body fluids, the agents responsible for acquired immunodeficiency syndrome (AIDS) or other sexually transmitted disease or hepatitis
17. Positive hepatitis B (HBV), hepatitis C (HCV) or HIV results
18. Subjects receiving prohibited medication as described in Section 4.2
19. Unwilling to avoid excessive sunlight exposure
20. Failure to satisfy the Investigator of fitness to participate for any other reason
21. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval within 10 days prior to administration or during the trial, and CYP2C8 substrates such as amiodarone, amodiaquine, paclitaxel, rosiglitazone, pioglitazone and repaglinide or CYP2C9 such as warfarin, tolbutamide, phenytoin, losartan, acenocoumarol within 1 month or six half lives (whichever is greater)
22. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
23. A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of BI 671800 in plasma over the time interval from 0 extrapolated to infinity) | Up to 24 hours after last drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of BI 671800 in plasma over the time interval from 0 to the time of the last quantifiable data point) | Up to 24 hours after drug administration
tmax (time from dosing to the maximum concentration of BI 671800 in plasma) | Up to 24 hours after drug administration
Cmax (the maximum concentration of BI 671800 in plasma) | Up to 24 hours after drug administration
λz (terminal rate constant in plasma) | Up to 24 hours after drug administration
t½ (terminal half-life of BI 671800 in plasma) | Up to 24 hours after drug administration
MRTpo (mean residence time of BI 671800 in the body after oral administration) | Up to 24 hours after drug administration
CL/F (apparent clearance of BI 671800 in the plasma after extravascular administration) | Up to 24 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | Up to 24 hours after drug administration
tlag (time to first quantifiable plasma concentration) | Up to 24 hours after drug administration
Number of patients with clinical significant findings in physical examination | Up to 10 days after last drug administration
Number of patients with clinical significant findings in vital signs | Up to 10 days after last drug administration
Number of patients with clinical significant findings in 12-lead electrocardiogram (ECG) | Up to 10 days after last drug administration
Number of patients with clinical significant findings in clinical laboratory tests | Up to 10 days after last drug administration
Number of patients with adverse events | Up to 10 days after last drug administration